CLINICAL TRIAL: NCT04034576
Title: The Impact of Session-introducing Mindfulness and Relaxation Interventions in Individual Training Psychotherapies for Children and Adolescents: a Randomized Controlled Trial.
Brief Title: Mindfulness and Relaxation Interventions in Individual Psychotherapies for Children and Adolescents
Acronym: MARS-CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Esslingen University of Applied Sciences (Other); Leibniz Institute for Research and Information in Education (Unknown)
Responsible Party: Principal Investigator, Julia Kalmar, Dr. Julia Kalmar, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARSCA
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hyperkinetic Disorder; Depressive Disorder; Anxiety Disorder
Keywords: Mindfulness-based intervention; Session-introducing interventions; Child and adolescent psychotherapy; Cognitive-behavioral therapy; Therapeutic alliance; Depressive disorder; Hyperkinetic disorder; Anxiety disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TAU + mindfulness intervention (Experimental): The mindfulness-based intervention consists of three five to ten minutes session-introducing interventions (mindful walking, body scan, breathing space). At the beginning of each of the 24 therapy sessions patients receive one of the three mindfulness interventions. Each intervention is instructed for four sessions consecutively and eight sessions in total. After completion of the mindfulness intervention, the regular therapy session begins.
  Interventions: Behavioral: Cognitive behavior therapy of trainee therapists
- TAU + relaxation intervention (Active Comparator): The relaxation interventions (progressive muscle relaxation (PMR), imagery journey, walking relaxation) are parallelized to the three mindfulness-based interventions. At the beginning of each of the 24 therapy sessions, patients receive one of the three relaxation interventions. Each intervention is instructed for four sessions consecutively and eight sessions in total. After completion of the relaxation intervention, the regular therapy session begins.
  Interventions: Behavioral: Cognitive behavior therapy of trainee therapists
- Treatment as usual (Other): Standard cognitive behavior therapy treatment, based on the individualized case conception of the trainee therapist, is conducted during the whole treatment sessions. No particular session-introductions are applied.
  Interventions: Behavioral: Cognitive behavior therapy of trainee therapists

INTERVENTIONS:
Behavioral: Cognitive behavior therapy of trainee therapists — In all three treatment arms, trainee therapists perform a cognitive behavior therapy (CBT) under conditions of the German health care system. This treatment is not a manualized intervention, but rather based on individualized treatment plans that have been developed together with expert supervisors during a five session diagnostic stage. Treatment duration is 24 sessions, while on average every fourth is supervized by an CBT expert therapist.

SUMMARY:
The study 'Mindfulness and Relaxation interventions in Individual Training Psychotherapies for Children and Adolescents' (MARS-CA) aims to examine the effects of short session-introducing interventions with mindfulness elements (SIIME) on juvenile patients' psychopathological symptomatology and therapeutic alliance at the beginning of the first 24 therapy sessions.

DETAILED DESCRIPTION:
Short session-introducing interventions with mindfulness elements (SIIME) shall be compared with session-introducing relaxation interventions (SIRI) and no session-introducing interventions (treatment as usual, (TAU)). Patients between 11 and 19 years and a primary diagnosis of hyperkinetic disorder, depressive disorder or anxiety disorder are invited to participate. Psychotherapy will be conducted by trainee therapists at a trainee outpatient clinic for children and adolescents. It is hypothesized that psychopathological symptomatology and therapeutic alliance improve more in the mindfulness condition than in the relaxation condition and TAU, and that mindfulness moderates the relationship between therapeutic alliance and psychopathological symptomatology stronger than the relaxation condition and TAU.

ELIGIBILITY:
Inclusion Criteria:

* A primary hyperkinetic disorder, depressive disorder or anxiety disorder diagnosis
* treatment at the Center for Psychological Psychotherapy, University of Heidelberg

Exclusion Criteria:

* age below 11 or above 19
* insufficient German language skills
* psychotic disorder
* acute suicidality

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Changes in Youth Self-Report 11-18 R (YSR 11-18 R) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  The YSR 11-18 R measures general symptom severity in patients. Eight different subscales are differentiated across 112 items: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, delinquent behavior, and aggressive behaviors. The three subscales anxious/depressed, withdrawn/depressed and somatic complaints are regarded as internalizing problems while the two subscales delinquent behavior and aggressive behavior are regarded as externalizing behavior. To calculate subscales as well as the total score corresponding items are summed. Items are rated on a 3-point Likert-scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true). Higher scores reflect higher symptom severity. T-scores are used to interpret and compare the results to the corresponding age and gender group.

SECONDARY OUTCOMES:
Therapeutic Alliance Scale for Children (FTB-KJ) | measured for 24 weeks on weekly basis at the end of each session (session duration is 50 minutes), starting on first treatment day
  The FTB-KJ is a self-report instrument to measure therapeutic alliance. It contains a patient and therapist perspective with 12 items rated on a four-step scale. In addition to the items of the FTB-KJ, a two-item short version of the Therapeutic Presence Inventory will be applied. Furthermore, two items will assess if patients and therapists perceive the session-introducing intervention positively or negatively.
Child and Adolescent Mindfulness Measure (CAMM) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  The CAMM is based on the Kentucky Inventory of Mindfulness Skilss (KIMS) and assesses the general development of mindfulness in patients.The measure includes ten items, rated on a five-step scale.
Self-compassion scale (SCS-D) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  To assess patients' and therapists' general development of self-compassion across the course of the study, we will apply the SCS and an adapted version of the SCS for children translated into German. It consists of 26 items and is rated on a five-step scale.
Diagnostic System for Mental Disorders in Childhood and Adolescence (DISYPS-III), problem scales of the ADHD self-rating scale (SBB-ADHS) Title: Patients' hyperkinetic disorder symptoms | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  To assess the patients' hyperkinetic disorder symptoms, we will apply the DISYPS-III SBB-ADHS, consisting of 20 items rated on a four-step scale.
Diagnostic System for Mental Disorders in Childhood and Adolescence (DISYPS-III), problem scales of the depression self-rating scale (SBB-DES) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  To assess depressive symptoms of the patients, we will apply the DISYPS-III SBB-DES. The problem scales of the SBB-DES consist of 29 items, rated on a four-step scale.
Diagnostic System for Mental Disorders in Childhood and Adolescence (DISYPS-III), problem scales of the anxiety self-rating scale (SBB-ANG) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  To assess anxiety symptoms of the patients, we will apply the DISYPS-III SBB-ANG. The problem scales of the SBB-ANG consist of 44 items, rated on a four-step scale.
Kentucky Inventory of Mindfulness Skills (KIMS-D) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  General development of mindfulness amongst therapists across the course of the study will be assessed by the German version of the KIMS. Ot consists of 39 items that are rated on a five-step scale

OTHER OUTCOMES:
Practice Quality-Mindfulness to patients (PQ-M) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  The six items of the PQ-M assess the perceived quality of mindfulness implementation operationalised as perseverance in (a) receptive (b) present-moment attention.
Credibility/Expectancy Questionnaire (CEQ) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  The questionnaire assesses treatment expectancy and rationale credibility in clinical outcome studies.
Heidelberg Inventory of Cognitive-Behavioral Interventions (HICBI) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  Assesses the application of specific therapeutic techniques
Therapist Presence Inventory (TPI) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  Assesses patients' and therapists' in-session therapeutic presence
Adherence scale (Ad-S) | on first treatment day, after 3 weeks, 10 weeks, 17 weeks, 24 weeks (in each case after a 50 minutes therapy session) and at a 6-month follow-up
  Was specifically designed to assess potential adherence effects in therapists and patients. It consists of 8 items in the patient version and 13 items in the therapist version. Patients rate five statements about how they perceived the session-introducing interventions (0 = not correct at all, 4 = true) and are asked whether and how often they practiced at home. The therapist version contains a list of 10 possible components for the session introduction (e.g. mindfulness intervention, review over the last session) that can be rated from 0 (not correct at all) to 4 (true). Also, therapists are asked to rate 3 statements about how they perceived the session introduction (0=not correct at all to 4= true).

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kalmar, Dr., Principal Investigator — Heidelberg University; Johannes Mander, PD Dr., Principal Investigator — Heidelberg University; Hinrich Bents, Dr., Study Director — Heidelberg University; Eva Vonderlin, Dr., Study Director — Heidelberg University; Thomas Heidenreich, Prof. Dr., Study Chair — University of Applied Sciences Esslingen; Sabina Pauen, Prof. Dr., Study Chair — Heidelberg University; Andreas Neubauer, Dr., Study Chair — Leibniz Institute for Research and Information in Education Frankfurt (Main)
Locations (1):
- Heidelberg University, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mander J, Blanck P, Neubauer AB, Kroger P, Fluckiger C, Lutz W, Barnow S, Bents H, Heidenreich T. Mindfulness and progressive muscle relaxation as standardized session-introduction in individual therapy: A randomized controlled trial. J Clin Psychol. 2019 Jan;75(1):21-45. doi: 10.1002/jclp.22695. Epub 2018 Oct 8. PMID 30295914
- [Derived] Kalmar J, Baumann I, Gruber E, Vonderlin E, Bents H, Neubauer AB, Heidenreich T, Mander J. The impact of session-introducing mindfulness and relaxation interventions in individual psychotherapy for children and adolescents: a randomized controlled trial (MARS-CA). Trials. 2022 Apr 11;23(1):291. doi: 10.1186/s13063-022-06212-0. PMID 35410284